CLINICAL TRIAL: NCT05394610
Title: A Confirmatory Investigation of the Effectiveness of Sana Treatment in Fibromyalgia
Brief Title: Effectiveness of the Sana Device on Fibromyalgia Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sana Health (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 850524
Record Dates: First submitted 2022-05-23; First posted 2022-05-27 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Fibromyalgia; Pain, Chronic; Quality of Life
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Double blind sham contolled
Who Masked: Participant, Investigator
Masking Description: Investigators and subjects will be blinded to the randomized arm assignment. Subjects will receive the Active Sana treatment OR Sham-controlled treament. The sham controlled device is physically identical to the active treatment, with pattern of lights and sound varying between the two.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Active Comparator): The Sana Device is an externally worn mask that physically contacts the skin of the face. The Sana Device delivers Audio Visual Stimulation (AVS) in the form of coordinated pulses of light (through closed eyelids) and sound at various frequencies. The device is externally communicating only. The Sana Device will be administered at least twice daily, with one treatment session being just prior to bedtime. Additional PRN sessions with the Sana device will be allowed at the subject's discretion.
  Interventions: Device: Sana Device
- Sham Arm (Sham Comparator): The sham treatment device was designed to copy the look and feel of the Sana therapy to a degree that it would be indistinguishable from the true treatment. The sham treatment delivers a series of Audio Visual Stimulation (AVS) in the form of pulses of light (through closed eyelids) and ound but should offer no therapeutic effect to the level of the Sana Device. The sham device will run on the same headset, use a matched intensity of light/audio and used on the same schedule as the Sana treatment.
  Interventions: Drug: Sana Device (Control)

INTERVENTIONS:
Device: Sana Device — Audio Visual Stimulation patterns intended to produce a therapeutic benefit.
  Arms: Active Treatment
Drug: Sana Device (Control) — A control device that mimics the physcial appearance of the Sana device.
  Arms: Sham Arm

SUMMARY:
This is study designed to confirm the effectiveness of the Sana Device in patients with pain due to fibromyalgia on quality of life as measured by the Fibromyalgia Impact Questionnaire Revised (FIQR). It is a two arm study in which subjects will be randomly assigned to either active device group or sham-controlled group.

ELIGIBILITY:
Inclusion Criteria:

* Willing to and capable of providing written informed consent prior to the conduct of any study-related procedures.
* Male or female, 18 to 65 years of age, inclusive.
* Have a history of experiencing fibromyalgia - like symptoms for a minimum of 36 months (3 years) prior to Screening.
* Subject must be in good physical health based on physical exams, vitals, and/or self-reporting. For subjects where there may not be sufficient recent medical records to document general good health the participant will be asked to self-report at the investigator's discretion.
* Any analgesic medications and medication dosages must be at approximately stable levels for at least 8 weeks prior to enrollment and remain steady throughout the study.
* A total score on the Generalized Anxiety Disorder 7-item scale (GAD-7) of 5 or above.
* A total score on the Patient Health Questionnaire 8-item (PHQ-8) of 5 or above.
* A total score on the STOP-Bang questionnaire of 3 or below.
* Willing and able to comply with the study requirements, complete study assessments, and participate at scheduled times for the duration of the Treatment Phase.
* Able to understand, speak and read English sufficient for the completion of study assessments.

Exclusion Criteria:

* Pregnant or lactating females as self-reported.
* History or presence of photo-sensitive epilepsy or other photo-sensitive conditions.
* History or presence of condition(s) that may affect balance, such as seizure disorders or vertigo.
* History of presence of condition (s) that meet the criteria for major depressive disorder (MDD), bipolar disorder, or any other personality disorders, at the discretion of the investigator.
* Presence of cancer pain, acute pain following injury or other severe pain not primarily associated with fibromyalgia, at discretion of the investigator.
* Surgery or trauma requiring rehabilitation within the last 12 weeks.
* Vision impairments that affect perception of light, color, or brightness in one or both eyes, and differences in visual perception between eyes.
* Deafness in one or both ears, perceived differences in hearing between ears, or tinnitus.
* Current ear or eye infection, untreated allergies, or acute illness that may affect eyes or hearing (e.g., due to congestion).
* Presence of inflammation or broken skin around the eyes in the area of the mask.
* Presence of narcolepsy or untreated sleep apnea or requiring treatment for sleep apnea such that use of device at bedtime will be interrupted, at discretion of the investigator.
* At the discretion of the Investigator, participation in any other clinical study in which medication(s) are being delivered or have used an investigational drug or device within the last 30 days.
* Any pending legal action that could prohibit participation or compliance in the study.
* Recent history of or current evidence of suicidal ideation or active suicidal behavior, based on medical history, at the discretion of the investigator.
* Significant medical conditions or other circumstances which, in the opinion of the investigator, would preclude compliance with the protocol, adequate cooperation in the study or obtaining informed consent, or may prevent the subject from safely participating in study.
* Employment by the investigator or the study site, with direct involvement in the proposed study or other studies under the direction of the investigator or study site, or a family member of an employee or of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in Fibromyalgia Symptoms | 6 weeks
  To confirm the superiority of the active arm over sham on changes in quality of life as measured by the Fibromyalgia Impact Questionnaire Revised (FIQR)

SECONDARY OUTCOMES:
Changes in Generalized Anxiety Symptoms | 6 weeks
  To confirm the superiority of the active arm over sham on generalized anxiety as measured by Generalized Anxiety Disorder 7-item (GAD-7)
Changes in Depression Symptoms | 6 weeks
  To confirm the superiority of the active arm over sham on depression sypmtoms as measured by the Patient Health Questionnaire-8 (PHQ-8)
Changes in Sleep Quality | 6 weeks
  To confirm superiority of the active arm over sham on sleep quality as measured by the PROMIS 4a Sleep Disturbance Scale (PR4A)
Changes in Pain | 6 weeks
  To confirm the superiority of the active arm over sham on reduction of pain as measured by the Pain Enjoyment General-Activity (PEG) scale
Perceived Change in Quality of Life | 6 weeks
  To examine the effect of the active arm on perceived change in quality of life as measured by the Patient Global Impression of Change (PGIC) scale

CONTACTS AND LOCATIONS:
Overall Officials: Martin Cheatle, PhD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No